CLINICAL TRIAL: NCT04427904
Title: Bupivacaine Versus Lidocaine Infiltration for Postoperative Pain in Thyroid Surgery: A Randomized Controlled Trial
Brief Title: Bupivacaine Versus Lidocaine Infiltration for Postoperative Pain in Thyroid Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Michael Xie, Resident Physician, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7336
Record Dates: First submitted 2020-05-26; First posted 2020-06-11 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Postoperative Pain; Thyroid Diseases; Anesthesia, Local
Keywords: Thyroidectomy; Bupivacaine; Lidocaine
MeSH Terms: conditions — Pain, Postoperative; Thyroid Diseases | interventions — Bupivacaine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine (Experimental): Bupivacaine 0.5% with 1:200 000 epinephrine. Total volume 10mL for local infiltration before neck incision.
  Interventions: Drug: Bupivacaine 0.5% with 1:200 000 epinephrine
- Lidocaine (Active Comparator): Lidocaine 2% with 1:100 000 epinephrine. Total volume 10mL for local infiltration before neck incision.
  Interventions: Drug: Lidocaine 2% with 1:100 000 epinephrine

INTERVENTIONS:
Drug: Bupivacaine 0.5% with 1:200 000 epinephrine — Bupivacaine 0.5% with 1:200 000 epinephrine. Total volume 10mL for local infiltration before neck incision.
  Other Names: Marcaine
  Arms: Bupivacaine
Drug: Lidocaine 2% with 1:100 000 epinephrine — Lidocaine 2% with 1:100 000 epinephrine. Total volume 10mL for local infiltration before neck incision.
  Other Names: Xylocaine
  Arms: Lidocaine

SUMMARY:
The purpose of this study is to compare the efficacy of Bupivicaine and Lidocaine for postoperative pain control in thyroid surgery.

DETAILED DESCRIPTION:
Patients planned for total thyroidectomy will be recruited for participation. After being informed about the study and potential risks, all patients giving written informed consent will be screened for eligibility for study entry. Patients that meet inclusion and exclusion criteria will be randomized via block randomization in a double blind fashion and a 1:1 ratio to surgical incision infiltration with Bupivacaine (0.5% with 1:200 000 epinephrine) or Lidocaine (2% with 1:100 000 epinephrine).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of thyroid disease (malignant tumors T1-T3/NX-N1a, benign tumors)
* Planned for thyroid surgery with midline neck incision (total thyroidectomy, completion thyroidectomy, with or without central neck dissection)
* Will be admitted for at least 12h postoperatively

Exclusion Criteria:

* Thyroid cancer staged as T4 (invasion, anaplastic) or requiring sternotomy
* Thyroid cancer staged as N1b (cervical, retropharyngeal, superior mediastinal nodal involvement)
* Previous ipsilateral thyroid surgery to operation side
* Previous total thyroidectomy or completion thyroidectomy
* History of neck radiation therapy
* Neck dissection beyond central neck (levels 1-5)
* Goiter extending beyond sternal notch (intrathoracic) or requiring sternotomy
* Surgery requiring extension of incision beyond 8 cm
* History of diabetes mellitus
* History of renal or liver disease
* History of narcotic abuse
* History of chronic pain medications use in past 6 months for any condition
* History of coagulation defect
* Allergy to Bupivacaine or Lidocaine

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | 30 minutes after surgery
  Patient reported postoperative pain reported on a 10cm pain visual analogue scale (VAS), minimum value of 0cm (no pain) and maximum value of 10cm (worst pain possible), lower VAS measurement represents better outcome
Postoperative Pain | 1 hour after surgery
  Patient reported postoperative pain reported on a 10cm pain visual analogue scale (VAS), minimum value of 0cm (no pain) and maximum value of 10cm (worst pain possible), lower VAS measurement represents better outcome
Postoperative Pain | 2 hours after surgery
  Patient reported postoperative pain reported on a 10cm pain visual analogue scale (VAS), minimum value of 0cm (no pain) and maximum value of 10cm (worst pain possible), lower VAS measurement represents better outcome
Postoperative Pain | 3 hours after surgery
  Patient reported postoperative pain reported on a 10cm pain visual analogue scale (VAS), minimum value of 0cm (no pain) and maximum value of 10cm (worst pain possible), lower VAS measurement represents better outcome
Postoperative Pain | 4 hours after surgery
  Patient reported postoperative pain reported on a 10cm pain visual analogue scale (VAS), minimum value of 0cm (no pain) and maximum value of 10cm (worst pain possible), lower VAS measurement represents better outcome
Postoperative Pain | 8 hours after surgery
  Patient reported postoperative pain reported on a 10cm pain visual analogue scale (VAS), minimum value of 0cm (no pain) and maximum value of 10cm (worst pain possible), lower VAS measurement represents better outcome
Postoperative Pain | 12 hours after surgery
  Patient reported postoperative pain reported on a 10cm pain visual analogue scale (VAS), minimum value of 0cm (no pain) and maximum value of 10cm (worst pain possible), lower VAS measurement represents better outcome

SECONDARY OUTCOMES:
First dose of additional postoperative analgesia | Up to 72 hours after surgery
  Time since completion of surgery when additional postoperative analgesia outside of standardized protocol was administered
Inpatient analgesia utilization | Up to 72 hours after surgery
  Quantity of standardized analgesia used during admission
Outpatient analgesia utilization | Up to 4 weeks after surgery
  Quantity of standardized analgesia used between discharge and 4 week outpatient follow up
Time to return of sensation | Up to 4 weeks after surgery
  Patient reported time to return of sensation at surgical site
Incidence of postoperative complications | 4 weeks
  Incidence of complications including bleeding, hematoma, surgical site infection, dehiscence, re-exploration, persistent paresthesia
Incidence of local anesthesia related adverse events | 4 weeks
  Incidence of adverse events including CNS (tinnitus, blurred vision, dizziness, tongue paresthesias, circumoral numbness, seizures, CNS depression) and cardiovascular (hear block, sinus bradycardia, sinus arrest, ventricular arrhythmias) events.
Postoperative pain | 1 week
  Patient reported postoperative pain reported on a 10cm pain visual analogue scale (VAS), minimum value of 0cm (no pain) and maximum value of 10cm (worst pain possible), lower VAS measurement represents better outcome
Postoperative pain | 2 week
  Patient reported postoperative pain reported on a 10cm pain visual analogue scale (VAS), minimum value of 0cm (no pain) and maximum value of 10cm (worst pain possible), lower VAS measurement represents better outcome
Postoperative pain | 4 week
  Patient reported postoperative pain reported on a 10cm pain visual analogue scale (VAS), minimum value of 0cm (no pain) and maximum value of 10cm (worst pain possible), lower VAS measurement represents better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Han Zhang, MD FRCSC, Principal Investigator — St. Joseph's Hospital Hamilton
Locations (1):
- St. Joeseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No